CLINICAL TRIAL: NCT01368926
Title: A Double-Blind, Randomized, Placebo-Controlled Study Evaluating the Pharmacokinetics, Safety and Tolerability of RO4917523 Conducted in 2 Phases: a Single-Dose, Cross-Over Administration to Healthy Japanese Subjects and a Multiple-Dose Administration to Healthy Japanese and Caucasian Subjects.
Brief Title: A Pharmacokinetic Study of RO4917523 in Healthy Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: BP25713
Record Dates: First submitted 2011-05-27; First posted 2011-06-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 2-chloro-4-(1-(4-fluorophenyl)-2,5-dimethyl-1H-imidazol-4-ylethynyl)pyridine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Part 1 (Experimental)
  Interventions: Drug: RO4917523; Drug: placebo
- Part 2 (Experimental)
  Interventions: Drug: RO4917523; Drug: placebo

INTERVENTIONS:
Drug: RO4917523 — single oral doses
  Arms: Part 1
Drug: RO4917523 — multiple oral doses
  Arms: Part 2
Drug: placebo — oral doses

SUMMARY:
This double-blind, randomized, placebo-controlled, 2-Part study will evaluate the pharmacokinetics and safety of RO4917523 in healthy Japanese and Caucasian volunteers. In Part 1, healthy Japanese volunteers will be randomized to receive 2 oral doses of either RO4917523 or placebo, with a washout period of 21 days between dosing. In Part 2, healthy Japanese and Caucasian volunteers will be randomized in cohorts to receive either RO4917523 or placebo orally daily for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese (Part 1 + 2) or Caucasian (Part 2) adults, 18- 50 years of age
* Japanese subjects must have Japanese parents and grandparents who were born in Japan
* Caucasian subjects must have 4 Caucasian grandparents
* Body mass index (BMI) 18.5 to 26 kg/m2, and a body weight of at least 45 kg
* Non-smoker for at least 90 days prior to dosing Day 1

Exclusion Criteria:

* Participation in a clinical trial with an investigational drug within 90 days prior to dosing Day 1. (Volunteers having participated in Part 1 will not be allowed to participate in Part 2 and vice versa)
* History or evidence of any clinically significant disease or disorder
* Pregnant or lactating women
* Positive for hepatitis B, hepatitis C or HIV
* Positive drug screen test, positive cotinine test and/or positive alcohol test
* Any confirmed significant allergic reactions to any drug, or multiple allergies in the judgement of the investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Part 1: Pharmacokinetics: Area under the concentration - time curve (AUC) (single/multiple oral dose in healthy Japanese subjects) | approximately 12 weeks
Part 2: Comparison of pharmacokinetics (area under the concentration - time curve [AUC]) between healthy Caucasian and Japanese subjects after 14 days of daily oral dosing | approximately 9 weeks
Safety: Incidence of adverse events in Japanese an Caucasian subjects | approximately 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- New York, New York, United States